CLINICAL TRIAL: NCT04552587
Title: A Mobile-Support Program to Facilitate Nutritional Caregiving in Head and Neck Cancer
Brief Title: The HEART Study (Healthy Eating and Recovery Together)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katherine Sterba, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0006621; R21CA215557-02 (NIH)
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Head and Neck Cancer; Survivorship; Nutrition Aspect of Cancer
Keywords: mHealth; Head and Neck Cancer; Survivorship; Caregiver
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEART (Experimental): Patients and caregivers will complete a HEART visit virtually or in person. The visit includes a needs assessment that generates a tailored care plan with messages, referrals and educational materials for discussion with a nurse. Caregivers will receive brief training about the HEART App and then use the App for 4 weeks with bi-weekly real-time prompts and feedback.
  Interventions: Behavioral: Heart APP

INTERVENTIONS:
Behavioral: Heart APP — The HEART intervention includes a care planning visit for patients and caregivers and an App for caregivers focused on nutrition, self-care and support.

SUMMARY:
Head and neck cancer survivors and their primary caregivers (N=25 dyads) will be enrolled to pilot test a nutrition support system with a care planning clinic visit and a caregiver mobile App. Participants will be asked to complete baseline and 6-week follow-up surveys. The clinic session (offered in person or remotely) will include a needs assessment and a tailored care plan with information, educational materials and referrals about participants' symptoms, behaviors, social concerns and caregiving tasks. After the visit, the program will provide an App for caregivers with follow-up resources and mobile support for one month.

DETAILED DESCRIPTION:
The long-term goal of this research is to improve physical, emotional and social post-treatment outcomes in head and neck cancer survivors and caregivers by implementing a nutrition-focused mobile-Support program to prepare and support caregivers after treatment.

Head and neck cancer survivors and their primary caregivers (N=25 dyads) will be recruited to a single-arm intervention study to evaluate the feasibility, acceptability and short-term effects of a nutrition-focused mobile support system. The intervention includes 1) a clinic visit (offered in-person or virtually) with a tablet-based needs assessment at the end of or after completing treatment which will generate 2) a tailored care plan with messages, educational materials and referrals mapped to survivor and caregiver-endorsed concerns and 3) a caregiver App with encouragement, reminders and tips delivered through messaging and peer videos. Participants will complete baseline and 6-week follow-up surveys.

ELIGIBILITY:
Patient Inclusion Criteria:

* 18 years and older
* Patients with stage I-IVB HNC of the upper aerodigestive tract (including lip/oral cavity, nasopharynx, salivary gland, oropharynx, hypopharynx, paranasal sinus, and larynx cancers and cutaneous cancers of the head and neck region)
* In the last two weeks of treatment to 3 months following completion of primary treatment (i.e., any combination of surgery, chemotherapy and radiation therapy) within the past 3 months
* Experienced nutritional challenges at the end of treatment as assessed in a 6-item screener

Patient Exclusion Criteria:

* head and neck cancer patients who do not undergo treatment
* Patients who do not read or understand English
* Patients who are cognitively impaired and cannot complete interviews, as judged by the referring health care provider
* Patients who do not have a smartphone for use in the study

Caregiver Inclusion Criteria:

* 18 years and older
* Provide care for a loved one with stage I-IVB head and neck cancer who has completed treatment

Caregiver Exclusion Criteria:

* Caregivers who do not read or understand English
* Caregivers who are cognitively impaired and cannot complete interviews, as judged by the referring health care provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sterba, PhD. MPH, Principal Investigator — Medical University of SC
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Head and neck cancer patients and caregivers were recruited at the end of radiation therapy.
Period: Overall Study
Arm/Group | HEART
Started | 50
Patients | 23
Caregivers | 23
Completed | 46 (N= 23 Patients, 23 Caregivers)
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | HEART
Number analyzed (Participants) | 46
Age, Continuous [Mean (Full Range); unit: years] — Population: 5 individuals who enrolled did not complete the study.
  years
    Caregivers: number analyzed (Participants) | 23
    Caregivers | 59 [21 to 83]
    Patients: number analyzed (Participants) | 23
    Patients | 63 [31 to 86]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 5 individuals who enrolled did not complete the study
  Participants
    Caregivers: number analyzed (Participants) | 23
    Caregivers: Female | 18
    Caregivers: Male | 5
    Patients: number analyzed (Participants) | 23
    Patients: Female | 7
    Patients: Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 5 individuals who enrolled did not complete the study
  Participants
    Caregiver: number analyzed (Participants) | 23
    Caregiver: Hispanic or Latino | 0
    Caregiver: Not Hispanic or Latino | 23
    Caregiver: Unknown or Not Reported | 0
    Patient: number analyzed (Participants) | 23
    Patient: Hispanic or Latino | 0
    Patient: Not Hispanic or Latino | 23
    Patient: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 5 individuals who enrolled in the study did not complete the study.
  Participants
    Caregivers: number analyzed (Participants) | 23
    Caregivers: American Indian or Alaska Native | 0
    Caregivers: Asian | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0
    Caregivers: Black or African American | 3
    Caregivers: White | 20
    Caregivers: More than one race | 0
    Caregivers: Unknown or Not Reported | 0
    Patients: number analyzed (Participants) | 23
    Patients: American Indian or Alaska Native | 0
    Patients: Asian | 0
    Patients: Native Hawaiian or Other Pacific Islander | 0
    Patients: Black or African American | 4
    Patients: White | 19
    Patients: More than one race | 0
    Patients: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting Patient-Caregiver Session and Care Plan Acceptability Criteria
Description: Investigator developed questionnaire investigating acceptability of session intervention and care plan. Items were rated on a 6-point descriptive scale from strongly disagree to strongly agree. Participants that meet criteria are those that chose moderately or strongly agree. Items included: Session made me feel prepared, care plan information was helpful emotionally, care plan was helpful practically, amount of information in care plan provided was appropriate, timing of session of session was appropriate.
Time Frame: 6 week follow-up visit
Measure: Number; unit: participants
Groups:
- HEART Patients; HEART Caregivers: Patients and caregivers will complete a HEART visit virtually or in person. The visit includes a needs assessment that generates a tailored care plan with messages, referrals and educational materials for discussion with a nurse. Caregivers will receive brief training about the HEART App and then use the App for 4 weeks with bi-weekly real-time prompts and feedback.
  Heart APP: The HEART intervention includes a care planning visit for patients and caregivers and an App for caregivers focused on nutrition, self-care and support
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
participants
  Session made me feel prepared | 18 | 18
  Care plan information was helpful emotionally | 17 | 15
  Care plan was helpful practically | 18 | 18
  Amount of information in the care plan provided was appropriate | 18 | 20
  Session timing was appropriate | 13 | 9

2. Primary Outcome: Intervention Delivery/ Fidelity
Description: Number of caregivers receiving all session content and delivery of the intervention as planned (intro to session, nurse care plan discussion, viewed nutritional support video, app training).
Time Frame: 6 week follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | HEART Caregivers
Number analyzed (Participants) | 23
Participants | 19

3. Primary Outcome: Intervention Reach
Description: Percentage of those recruited who completed baseline and 6 week follow up surveys and the intervention session.
Time Frame: Baseline and 6 week follow up visit
Population: 50 enrolled, 4 lost to follow up
Measure: Count of Participants; unit: Participants
Groups:
- HEART Total: Patients and caregivers will complete a HEART visit virtually or in person. The visit includes a needs assessment that generates a tailored care plan with messages, referrals and educational materials for discussion with a nurse. Caregivers will receive brief training about the HEART App and then use the App for 4 weeks with bi-weekly real-time prompts and feedback.
  Heart APP: The HEART intervention includes a care planning visit for patients and caregivers and an App for caregivers focused on nutrition, self-care and support.
Arm/Group | HEART Total
Number analyzed (Participants) | 50
Participants | 46

4. Secondary Outcome: Ease of Use/System Usability
Description: System Usability Scale (SUS) - The SUS consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Scores range from 0-100, with higher scores indicating better usability.
Time Frame: 6 week follow up visit only (no baseline comparison)
Population: System Usability Scale only measured in Caregivers.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HEART Caregivers
Number analyzed (Participants) | 23
score on a scale | 76 [20 to 98]

5. Secondary Outcome: Mean Score of Unmet Needs
Description: 30-item Cancer Survivors/Partners Unmet Needs instruments (CaSUN/ CaSPUN). Needs were endorsed on a yes/no basis, with a range of 0-30 total endorsed needs. A higher score indicates more endorsed needs. Average number of needs is reported.
Time Frame: Baseline and 6 week follow up visit
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
score on a scale
  Baseline endorsed needs | 9.5 [5.8 to 13.2] | 8.6 [5.5 to 11.7]
  6 week follow up visit endorsed needs | 8.9 [5.4 to 12.5] | 7.5 [4.1 to 10.9]
  Change from baseline to 6 week follow up visit | -0.6 [-2.7 to 1.6] | -1.0 [-3.7 to 1.6]

6. Secondary Outcome: PROMIS Depression- Short Form (SF) v1.0 Form 8A
Description: PROMIS Depression- SF v1.0 form 8A is an 8-item Patient-Reported Outcomes Measure Information System (PROMIS) short-form instrument. Respondents are asked how often in the past 7 days they have experienced specific depression symptoms, using a 5-point ordinal rating scale of "Never," "Rarely," "Sometimes," "Often," and "Always" whereby a higher score indicates higher depression. Raw score totals are converted to an item response theory-based T-scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10 with a range of 38.2 to 81.3. Therefore, a person with a T-score of 40 is one SD below the mean. A decrease in change from baseline to 6 week followup indicates reduced depression.
Time Frame: Baseline and 6 week follow-up visit
Measure: Mean (Full Range); unit: T-Score
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
T-Score
  Baseline | 51.2 [47.2 to 55.1] | 51.1 [47.3 to 54.9]
  6 week follow up visit | 48.0 [44.0 to 52.0] | 49.6 [45.8 to 53.4]
  Change from baseline to 6 week follow up visit | -3.2 [-6.0 to -0.3] | -1.5 [-4.7 to 1.8]

7. Secondary Outcome: Mean Score of Survivorship Readiness/Caregiver Preparedness
Description: The 11-item Preparing for Life As a New Survivor (PLANS) Knowledge Subscale, developed at the University of Michigan, is utilized to evaluate survivor and caregiver (1) knowledge of diagnosis, treatment and side effects, and (2) communication with the cancer team regarding diagnosis, treatment and side effects and 3) preparedness for what to expect over the next year. Items are rated on a 6-point scale where: strongly disagree=1, moderately disagree =2, slightly disagree=3, slightly agree= 4, moderately agree=5 and strongly agree=6. Items were averaged, with a range of 1-6 with higher scores indicating higher levels of agreement.
Time Frame: Baseline and 6 week follow-up visit
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
score on a scale
  Baseline | 4.5 [4.2 to 4.9] | 4.6 [4.1 to 5.0]
  6 week follow up visit | 4.6 [4.2 to 5.1] | 4.5 [4.0 to 5.0]
  Change from baseline to 6 weeks follow up | 0.1 [-0.3 to 0.4] | -0.1 [-0.4 to 0.3]

8. Secondary Outcome: Mean Score of Self-Efficacy
Description: Based on the National Cancer Institute Follow-up Care Use Among Survivors (FOCUS) survey, two questions were asked: "How confident are you that you can get advice or information related to your/your loved one's cancer if you needed at this time?" and "How confident are you that you can (assist your loved one to) keep to the follow-up care schedule recommended by your doctors?" Participants rated items on a 5-point Likert scale where 0="Not at all confident" to 4= "Completely confident." Scores were averaged for each question, whereby higher scores indicated higher level of confidence. Change from baseline to 6 week follow up is also reported. Negative change indicates decline in self-efficacy.
Time Frame: Baseline and 6 week follow-up visit
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
score on a scale
  Baseline- Self Efficacy: confidence in obtaining cancer related advice | 3.3 [2.9 to 3.6] | 3.0 [2.5 to 3.5]
  6 week f/u Self Efficacy: confidence in obtaining cancer related advice/adhering to follow up care | 3.2 [2.8 to 3.6] | 2.8 [2.3 to 3.3]
  Change- Self Efficacy: confidence in obtaining cancer related advice/adhering to follow up care | -0.1 [-0.5 to 0.4] | -0.2 [-0.8 to 0.4]
  Baseline- Self Efficacy: adhering to recommended follow up care | 3.6 [3.4 to 3.6] | 3.3 [3.0 to 3.7]
  6 week f/u visit- Self Efficacy: adhering to recommended follow up care | 3.6 [3.3 to 3.8] | 3.4 [3.1 to 3.7]
  Change - Self Efficacy: adhering to recommended follow up care | 0.0 [-0.2 to 0.2] | 0.1 [-0.4 to 0.5]

9. Secondary Outcome: Mean Score of Dyadic Coping/ Dyadic Efficacy
Description: Dyadic Coping was measured using a 5-item cancer-specific subscale version of the Dyadic Coping Inventory. Items are rated on a 5-point scale from 1 ("never") to 5 ("always"). Scores were averaged with a higher score indicating a better outcome. A decrease in change between baseline and 6 week followup visit indicates worsening outcome over time.
  Dyadic Efficacy is an investigator developed 1-item question "How confident are you that you and your loved one can work together as a team to manage the cancer-related problems that come up?" Item was answered on a scale of 0 ("not at all confident") to 10 ("extremely confident"), with average score reported. A decrease in change between baseline and 6 week followup visit indicates worsening, where as an increase in change indicates improvement.
Time Frame: Baseline and 6 week follow-up visit
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
score on a scale
  Dyadic Coping: Baseline | 4.3 [4.0 to 4.7] | 4.1 [3.6 to 4.5]
  Dyadic Coping: 6 week follow up visit | 4.2 [3.8 to 4.6] | 4.1 [3.6 to 4.5]
  Dyadic Coping: Change from baseline to 6 week follow up | -0.2 [-0.4 to 0.1] | 0.0 [-0.4 to 0.4]
  Dyadic Efficacy: Baseline | 9.0 [7.9 to 10.0] | 8.2 [7.4 to 9.0]
  Dyadic Efficacy: 6 week follow up visit | 8.3 [7.3 to 9.3] | 8.6 [7.8 to 9.4]
  Dyadic Efficacy: Change from baseline to 6 week follow up | -0.6 [-1.3 to 0.1] | 0.4 [-0.3 to 1.2]

10. Secondary Outcome: Health-Related Quality-of-Life (PROMIS Scale v1.2 - Global Health)
Description: PROMIS Scale v1.2 - Global Health short form consists of 10 items that assess overall perceived quality of life and five general domains of health and functioning including overall physical health, mental health, social health, pain, and fatigue. Scoring uses a 5-point Likert scale with the response scores reversed (5=None to 1=Very severe) so that higher scores for responses always indicate better health. Raw scores are summed and converted to a T-score (mean score of 50, SD ± 10), Therefore a person with a T-score of 40 is one SD below the mean. A decrease in the change from baseline to 6 week follow up indicates worsening quality of life, whereas an increase indicates improvement.
Time Frame: Baseline and 6 week follow-up visit
Measure: Mean (Full Range); unit: T-Score
Groups:
- Patient HRQOL Mental Scores: Patient HRQOL Mental scores Patients and caregivers will complete a HEART visit virtually or in person. The visit includes a needs assessment that generates a tailored care plan with messages, referrals and educational materials for discussion with a nurse. Caregivers will receive brief training about the HEART App and then use the App for 4 weeks with bi-weekly real-time prompts and feedback.
  Heart APP: The HEART intervention includes a care planning visit for patients and caregivers and an App for caregivers focused on nutrition, self-care and support
- Caregiver HRQOL Mental Scores: Caregiver HRQOL Mental scores
  Patients and caregivers will complete a HEART visit virtually or in person. The visit includes a needs assessment that generates a tailored care plan with messages, referrals and educational materials for discussion with a nurse. Caregivers will receive brief training about the HEART App and then use the App for 4 weeks with bi-weekly real-time prompts and feedback.
  Heart APP: The HEART intervention includes a care planning visit for patients and caregivers and an App for caregivers focused on nutrition, self-care and support
- Patient HRQOL Physical Scores: Patient HRQOL Physical scores
  Patients and caregivers will complete a HEART visit virtually or in person. The visit includes a needs assessment that generates a tailored care plan with messages, referrals and educational materials for discussion with a nurse. Caregivers will receive brief training about the HEART App and then use the App for 4 weeks with bi-weekly real-time prompts and feedback.
  Heart APP: The HEART intervention includes a care planning visit for patients and caregivers and an App for caregivers focused on nutrition, self-care and support
- Caregiver HRQOL Physical Scores: Caregiver HRQOL Physical scores
  Patients and caregivers will complete a HEART visit virtually or in person. The visit includes a needs assessment that generates a tailored care plan with messages, referrals and educational materials for discussion with a nurse. Caregivers will receive brief training about the HEART App and then use the App for 4 weeks with bi-weekly real-time prompts and feedback.
  Heart APP: The HEART intervention includes a care planning visit for patients and caregivers and an App for caregivers focused on nutrition, self-care and support
Arm/Group | Patient HRQOL Mental Scores | Caregiver HRQOL Mental Scores | Patient HRQOL Physical Scores | Caregiver HRQOL Physical Scores
Number analyzed (Participants) | 23 | 23 | 23 | 23
T-Score
  Baseline | 47.7 [43.5 to 51.8] | 49.0 [45.4 to 52.6] | 42.4 [39.5 to 45.2] | 50.4 [47.8 to 53.1]
  6 week follow up visit | 46.6 [43.8 to 49.5] | 48.5 [44.2 to 52.7] | 44.6 [41.4 to 47.7] | 50.4 [47.5 to 53.3]
  Change from baseline to 6 week follow up visit | -1.0 [-4.0 to 1.9] | -0.5 [-3.5 to 2.5] | 2.2 [0.04 to 4.4] | -0.05 [-1.8 to 1.7]

11. Secondary Outcome: Caregiver Burden
Description: 4-item screening version of the Zarit Burden Interview is a self-report measure of caregiver burden. Caregivers rate each item on a 5-point Likert scale (0=never, 4= nearly always). Higher scores indicate greater caregiver distress. Total score range: 0 to 16, ≥ 8: high burden. An increase in change from baseline to 6 week follow up visit indicates increased caregiver distress.
Time Frame: Baseline and 6 week follow up visit
Population: Change in mean score from baseline to six weeks measured in caregivers only
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | HEART Caregivers
Number analyzed (Participants) | 23
units on a scale
  Baseline | 1.8 [1.5 to 2.1]
  6 Week follow up visit | 1.9 [1.6 to 2.3]
  Change from baseline to 6 week follow up visit | 0.1 [-0.1 to 0.4]
Statistical Analysis 1: Comparison: HEART Caregivers; We compared change from baseline to follow up in our single group of caregivers; Test type: Superiority; p = 0.23, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Ease of Mobile App Use/User Engagement
Description: Number of weekly prompt responses missed out of 184 total expected (23 caregivers given 2 prompts per week for 4 weeks).
Time Frame: 4 weeks during app use
Population: Measured in Caregivers only. (23 caregivers given 2 prompts per week for 4 weeks= 184 prompts).
Measure: Number; unit: number of missed prompts
Units Other Than Participants: prompts
Arm/Group | HEART Caregivers
Number analyzed (Participants) | 23
Number analyzed (prompts) | 184
number of missed prompts | 70

13. Secondary Outcome: Number of Participants With Care Plan Use Endpoints
Description: Number of participants of use of care plan after session, including patient and caregiver report of "Referred to Care Plan again," "Used Care Plan," "Used educational materials," and "Shared Care Plan with others."
Time Frame: 6 week follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
Participants
  Referred to Care plan again | 17 | 20
  Used Care Plan | 10 | 8
  Used educational materials | 10 | 16
  Shared Care Plan with others | 7 | 4

14. Secondary Outcome: Percentage of Participants Rating App Satisfaction/ Perceived Importance
Description: Ratings of satisfaction with app and prompts on a 6 point descriptive rating scale ranging from strongly agree to strongly disagree. Measurements reported below are count of participants who moderately or strongly agreed with individual prompts.
Time Frame: 6 week follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
Participants
  App support received helped you provide care for your loved one | 17 | 13
  App support was helpful emotionally | 15 | 11
  App provided practical tips | 10 | 12
  Amount of app information was appropriate | 15 | 16

15. Secondary Outcome: Process Monitoring Data
Description: Resources needed: Session length overall, length of nursing portion of session, length of app training- number of minutes
Time Frame: After session completion
Measure: Mean (Full Range); unit: minutes
Arm/Group | HEART Caregivers
Number analyzed (Participants) | 23
minutes
  Length of full session | 51 [31 to 80]
  Length of nursing visit (within full session) | 13 [3 to 30]
  Length of App Training | 12 [7 to 35]

16. Secondary Outcome: Change From Baseline in Nutritional Status Scale
Description: Investigator-developed 1 item: "During the past two weeks, how satisfied have you been with your nutritional status (from Extremely satisfied (1) to Not at all satisfied (5))?"
Time Frame: Baseline and 6 week follow up visit
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
score on a scale
  Baseline | 3.5 [3.0 to 4.0] | 3.3 [2.7 to 3.9]
  6 week follow up visit | 3.0 [2.6 to 3.5] | 2.5 [2.1 to 3.0]
  Change from baseline to 6 week follow up visit | -0.5 [-1.0 to 0] | -0.8 [-1.4 to -0.2]

17. Secondary Outcome: Change From Baseline in Symptom Distress/Symptom Management
Description: Adapted Symptom Distress Scale 1 item scaled to assess how distressing symptoms are to participant. 0= not at all distressing, 10= extremely distressing
  1 item to assess patient and caregiver perceptions concerning patient ability to manage symptoms. 0= can manage extremely well, 10= cannot manage at all
Time Frame: Baseline and 6 week follow up visit
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
score on a scale
  Symptom Distress: Baseline | 4.6 [3.4 to 5.8] | 5.6 [4.2 to 6.9]
  Symptom Distress: 6 week follow up | 4.2 [2.8 to 5.6] | 4.3 [3.0 to 5.6]
  Symptom Distress: Baseline to 6 week follow up visit | -0.4 [-1.8 to 1.0] | -1.3 [-2.7 to 0.2]
  Symptom Management: Baseline | 2.5 [1.3 to 3.6] | 3.7 [2.6 to 4.9]
  Symptom Management: 6 week follow up | 2.7 [1.7 to 4.0] | 2.6 [1.5 to 3.7]
  Symptom Management: Baseline to 6 week follow up visit | 0.2 [-1.1 to 1.6] | -1.2 [-2.3 to 0]

18. Secondary Outcome: Change From Baseline in Emotional Support
Description: PROMIS Short Form v2.0 - Emotional Support - 4a is a 4-item questionnaire. Item banks (currently adults only) assess perceived feelings of being cared for and valued as a person; having confidant relationships. PROMIS instruments are scored using item-level calibrations. Each question usually has five response options ranging in value from one to five. Raw scores are the sum of values of the response to each question then rescaled to to a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean.
Time Frame: Baseline and 6 week follow up visit
Measure: Mean (Full Range); unit: T-Score
Arm/Group | HEART Patients | HEART Caregivers
Number analyzed (Participants) | 23 | 23
T-Score
  Baseline | 56.0 [52.2 to 59.8] | 52.0 [48.1 to 55.8]
  6 week follow up visit | 55.7 [52.5 to 58.9] | 52.8 [49.5 to 56.0]
  Change from baseline to 6 week follow up visit | -0.3 [-2.6 to 1.9] | 0.8 [-2.7 to 4.4]

19. Secondary Outcome: Change From Baseline in Symptom Severity
Description: MD Anderson Symptom Inventory (MDASI) Head and Neck Module- Includes 13 core items and an additional 9 head and neck cancer module items which calculates a total score of symptom severity. The MDASI assesses the severity of symptoms at their worst in the last 24 hours on a 0-10 Numeric Rating Scale, with 0 being "not present" and 10 being "as bad as you can imagine." Core items and module symptom items are averaged into a mean module severity. A higher score always indicates an increase in severity. A decrease in change from baseline to 6 week follow up indicates improvement of symptoms.
Time Frame: Baseline and 6 week follow up visit
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HEART Patients
Number analyzed (Participants) | 23
score on a scale
  Baseline | 3.0 [2.4 to 3.7]
  6 week follow up visit | 2.0 [1.3 to 2.8]
  Change from baseline to 6 week follow up visit | -1.0 [-1.6 to -0.4]

ADVERSE EVENTS:
Time Frame: Baseline to 6 weeks followup
Arm/Group | HEART Patients | HEART Caregivers
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT04552587/Prot_SAP_001.pdf
  • Informed Consent Form: Patient Consent (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT04552587/ICF_002.pdf
  • Informed Consent Form: Caregiver consent (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT04552587/ICF_003.pdf